CLINICAL TRIAL: NCT04507386
Title: Reducing Sedentary Time in Patients With Mild Cognitive Impairment: The Take a STAND for Health Study TS4H-MCI
Brief Title: Reducing Sedentary Time in Patients With Mild Cognitive Impairment: The Take a STAND for Health Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Take a STAND for Health MCI
Record Dates: First submitted 2020-07-30; First posted 2020-08-11 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Health

STUDY DESIGN:
Intervention Model Description: A 4-month parallel-group randomised controlled trial will be performed, in which patients with mild cognitive impairment will be assessed at baseline (PRE) and after 4 months (POST). Moreover, a sub-sample of patients will perform a randomised crossover trial at baseline (PRE). Patients will complete three experimental sessions in a random manner, as follows: Prolonged sitting (SIT), in which participants engaged in prolonged sitting throughout an 5-h period and were instructed to minimize excessive movement; Exercise followed by prolonged sitting (EX), in which participants performed a 30-min moderate-to-vigorous exercise bout on a treadmill, subsequently, participants engaged in prolonged sitting as described for SIT; Light-intensity breaks (BR), in which participants completed a 3-min bout of light-intensity walking every 30 min of sitting throughout the experimental period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Take a STAND for health (Experimental): A newly developed personalized intervention focused on replacing sedentary time with light-(or very light-) intensity physical activity
  Interventions: Behavioral: Take a STAND for health
- Control (No Intervention): The control group will receive regular medical care and advice on healthy lifestyle, including physical activity and healthy eating recommendations

INTERVENTIONS:
Behavioral: Take a STAND for health — The Take a STAND for health is a newly developed 4-month goal-setting intervention aimed at reducing sedentary behavior
  Arms: Take a STAND for health

SUMMARY:
This research program aims to comprehensively investigate the clinical, physiological, metabolic, and molecular effects of reducing sedentary behavior in patients with mild cognitive impairment. A 4-month parallel-group randomized controlled trial will be conducted aiming to investigate the feasibility and efficacy of a newly developed personalized intervention focused on replacing sedentary time with light-(or very light-) intensity physical activity in patients with mild cognitive impairment. Additionally, a sub-sample of patients will complete a randomised cross-over study aiming to unravel potential mechanisms underlying the metabolic, physiological and molecular effects of breaking up sedentary time with light-intensity physical activity versus carrying out the minimum amount of daily exercise at once and then remaining sedentary versus simply remaining sedentary throughout all sessions, in a well-controlled laboratorial condition.

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged and older adults with mild cognitive impairment confirmed by a team of neurologists from the CEREDIC HC-FMUSP

Exclusion Criteria:

* Patients who spend less than 8 hours per day in sedentary time
* Patients who are physically active (more than 150 min/week of moderate physical activity, or more than 75 min/week of vigorous activity)
* Patients who are functional illiterates
* Patients with history or clinical diagnosis of neurological diseases
* Patients with severe psychiatric symptoms
* Patients taking antidepressants
* Patients with visual and/or hearing impairments that prevent participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Sedentary behaviour assessed by ActivPAL™ | 4 months

SECONDARY OUTCOMES:
Physical activity levels assessed by ActiGraph GT3X® | 4 months
Cognitive performance assessed by the Montreal Cognitive Assessment (MoCA) | 4 months
  Questionnaire to be completed by the patient. Final score 0 to 30, lower scores indicate worse cognitive performance
Cognitive decline assessed by the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE) | 4 months
  Questionnaire to be completed by the caregiver. 26 Likert scale questions. Higher scores indicate worse cognitive performance
Subjective memory complaints assessed by the Memory Complaint Scale (MCS) | 4 months
  Questionnaire to be completed by the patient and the caregiver. Final scores classify memory complaints as absent, mild, moderate or accentuated
Functional impairments in activities of daily living assessed by the Functional Activities Questionnaire (FAQ) | 4 months
  Questionnaire to be completed by the caregiver. Final score 0 to 30, higher scores indicate greater functional dependency
Anxiety symptoms assessed by the Geriatric Anxiety Inventory (GAI) | 4 months
  Questionnaire to be completed by the patient. Final score 0 to 20, higher scores indicate greater anxiety symptoms
Depression symptoms assessed by the Geriatric Depression Scale (GDS-15) | 4 months
  Questionnaire to be completed by the patient. Final score 0 to 15, higher scores indicate greater depression symptoms
Neurocognitive assessment assessed by the Cogstate Research™ (Cogstate, Melbourne, AUS) | 4 months
  Reliable online system that assesses verbal learning capacity, executive function, processing speed, attention capacity, reaction time, and operational memory. Final score will be generated automatically by the system
Magnetic resonance imaging using the Philips ACHIEVA 3.0 Tesla | 4 months
  The following sequences will be obtained: 1 - sagittal 3D T1; 2 - axial T2 fast spin echo (FSE); 3 - axial fluid-attenuated inversion recovery (FLAIR); 4 - coronal T2 spectral presaturation with inversion recovery (SPIR); 5 - coronal T2 aligned with hippocampus; 6 - SENSE diffusion
Positron emission computed tomography with 18F-fluordesoxyglucose (PET-18FDG) using the Biograph, CTI/Siemens, Knowville, EUA | 4 months
  Tomographic sections will be acquired for 15 minutes with a 256x256 matrix, zoom 2.5, resulting in pixels of size 1.04 mm (voxel of 1.04 mm3). The images will be reconstructed using the ordered subset expectation maximization (OSEM) iterative method, with six iterations and 16 subsets, and smoothed with a 5 mm Gaussian filter. The data will be corrected for scattering, attenuation and decay
Assessment of cerebrovascular reactivity to CO2 inhalation | 4 months
  Patients will wear a mask connected to a unidirectional valve with a Douglas bag (with 5% CO2). Evaluations will include: partial pressure of carbon dioxide at the end of expiration (PetO2, PetCO2) (Metalyzer model III b/breath-by-breath, CORTEX, Germany) and O2 saturation (SpO2; Nellcor, Medtronic Corporation, USA). Blood flow and diameter of the internal carotid artery will be assessed using a Doppler ultrasound (Logiq E, General Electric, Milwaukee, USA) connected to a linear transducer (12L-RS - 5.0-13.0 MHz). Cerebrovascular reactivity will be assessed by responses of arterial diameter, blood flow and shear rate to CO2 inhalation (reactivity = peak - baseline). A software with automatic detection of the artery walls will be used (Cardiovascular Suite, Quipu®, Pisa, Italy). Blood flow will be calculated (Flow = Vm x πr2 x 60). The shear rate will be calculated using the following formula: Shear rate = 8 x Vm / diameter
Muscle functional assessed by the Timed Stands Test and the Timed Up-and-Go Test | 4 months
  Test results will be combined to report muscle function
Handgrip strength assessed by a hand dynamometer | 4 months
  Patient will have three 5-second trials, with 1-minute interval between trials. Best score will be considered handgrip strength
Blood pressure | 4 months
Fatigue severity assessed by the Fatigue Severity Scale (FSS) | 4 months
Physical and mental aspects of fatigue assessed by the Chalder Fatigue Scale (CFS) | 4 months
Subjective sleep quality assessed by the Pittsburgh Sleep Quality Index (PSQI) | 4 months
Daytime sleepiness assessed by the Epworth Sleepiness Scale (ESS) | 4 months
Quality of life assessed by the SF-36 (Medical Outcomes Study 36 - Short-Form Health Survey) | 4 months
Food consumption | 4 months
  24-hour dietary recalls
Insulin sensitivity | 4 months
  Fasting serum concentrations of glucose, insulin
Lipid profile | 4 months
  Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Inflammatory cytokines | 4 months
  pro- and anti-inflammatory cytokines: IL-1, IL-1ra, IL-6, IL-10 e TNF-alpha
Genetic profile for Alzheimer's disease | 4 months
  Genotyping of apolipoprotein E (ApoE)
Oral glucose tolerance test | 4 months
  Fasting, 30, 60, 90, and 120 minutes

IPD SHARING:
Plan to Share IPD: No